CLINICAL TRIAL: NCT05553691
Title: An Open-Label Study Investigating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics & Exploratory Efficacy of Intravenous SPL026 Drug Product (DMT Fumarate) Alone or in Combination With SSRIs in Patients With Major Depressive Disorder
Brief Title: SPL026 With or Without SSRIs in Participants With MDD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Small Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT026_004; 2022-001767-27 (EudraCT Number)
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD; Depression; SSRI; N,N-dimethyltryptamine; DMT
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Intervention Model Description: Test Cohort of patients already taking an SSRI for their depression, compared to the Control Cohort who are not already taking an SSRI. All patients will receive SPL026
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Cohort (Experimental): Patients who are currently taking an SSRI that is not effective in fully relieving their depression (prescribed outside of study). Patients will be administered a single dose of SPL026 by intravenous infusion.
  Interventions: Drug: SPL026
- Control Cohort (Experimental): Patients who are not currently taking any pharmacological treatment for their depression. Patients will be administered a single dose of SPL026 by intravenous infusion.
  Interventions: Drug: SPL026

INTERVENTIONS:
Drug: SPL026 — Intravenous
  Other Names: N,N-dimethyltryptamine; DMT

SUMMARY:
The main aim of the study is to test the safety and tolerability of single doses of SPL026 (N,N-dimethyltryptamine [DMT] fumarate, a psychedelic tryptamine) in patients currently taking a selective serotonin reuptake inhibitor (SSRI) for their depression, but for whom the SSRI is not fully relieving their depression.

ELIGIBILITY:
Inclusion Criteria:

* MDD diagnosis
* Previously tried at least one approved method of treatment for their depression
* No monoamine oxidase-inhibitor class antidepressants for at least 3 months
* Deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, laboratory tests of blood and urine
* No psychedelic drug use in the 6 months before dosing until the end of the study
* Willing to follow the contraception requirements of the trial
* Willing to be contacted by email and video call, and have online access
* Able to give fully informed written consent
* Test Cohort only: currently on a stable dose of an unspecified single SSRI alone and not in combination with any other psychiatric medications, for at least 6 weeks prior to Screening with no intention of making any changes
* Control Cohort only: no antidepressant medication for 6 months before dosing

Exclusion Criteria:

* Substance use disorder
* Current or clinically relevant history of a psychotic disorder, or first-degree relatives with a clinically relevant history of a psychotic disorder
* Significant history of mania
* Significant risk of suicide
* Clinically relevant abnormal findings at the screening assessment
* Blood pressure, heart rate, or QTcF outside the acceptable ranges
* Acute or chronic illness (other than MDD) or infection
* Clinically relevant abnormal medical history or concurrent medical condition (other than MDD)
* Use of any serotonergic psychedelics within 6 months prior to dosing
* Patients of child-bearing potential who are pregnant or lactating, or who are sexually active and not using a reliable method of contraception
* History of a severe adverse reaction to any drug or sensitivity to serotonergic psychedelic drugs
* Use of over-the-counter or prescribed medication (excluding oral contraceptives, hormone replacement therapy and SSRIs [Test Cohort only]) within previous 28 day before dose of trial medication; or paracetamol or ibuprofen within 4 hours prior to dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability: Adverse Events | Screening to End-of-Study Follow-up (Day 29)
  Adverse events (AEs)
Safety & tolerability: Lab biochemistry | Screening, Day -1 and Day 1
  Values of potential clinical importance
Safety & tolerability: Vital signs - Heart Rate | Screening to Day 2
  Heart rate
Safety & tolerability: Vital signs - Blood pressure | Screening to Day 2
  Blood pressure
Safety & tolerability: Vital signs - Temperature | Screening to Day 2
  Temperature
Safety & tolerability: Electrocardiogram | Screening to Day 2
  QTcX intervals
Safety & tolerability: Suicidal Ideation | Screening to End-of-Study Follow-up (Day 29)
  Columbia-Suicide Severity Rating Scale

SECONDARY OUTCOMES:
Evaluation of plasma levels of DMT | 2, 5, 7, 10, 11, 13, 15, 30, 60, 120, 240 minutes post-dose
  Pharmacokinetic parameter calculation in the Test Cohort compared to the Control Cohort
Mystical Experience Questionnaire (MEQ) | Day 1 (dosing day)
  MEQ in the Test Cohort compared to the Control Cohort
Challenging Experience Questionnaire (CEQ) | Day 1 (dosing day)
  CEQ in the Test Cohort compared to the Control Cohort
Ruminative Responses Scale (RRS) | Day -1 and Day 29
  RRS in the Test Cohort compared to the Control Cohort
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Day -1, Day 15 and Day 29
  WEMWBS in the Test Cohort compared to the Control Cohort

OTHER OUTCOMES:
Exploratory efficacy: Montgomery-Åsberg Depression Rating Scale (MADRS) | Day -1, Day 8, Day 15 and Day 29
  MADRS in the Test Cohort compared to the Control Cohort

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Devlin, MD, Principal Investigator — MAC Clinical Research; Neel Bhatt, MD, Principal Investigator — MAC Clinical Research
Locations (2):
- United Kingdom (2):
  - Mac Clinical Research, Manchester, Greater Manchester
  - MAC Clinical Research, Liverpool, Prescot

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted Clinical Study Report Synopsis — https://www.isrctn.com/ISRCTN10974027